CLINICAL TRIAL: NCT06367387
Title: Pain Self-Management and Patient-Oriented Dosing for Pain and Retention in Office-based Addiction Treatment: a Randomized Trial
Brief Title: Pain Self-Management and Patient-Oriented Dosing for Pain and in Retention Opioid Treatment
Acronym: TREETOP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erin Winstanley (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Erin Winstanley, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23080191; RM1DA055311 (NIH)
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder; Chronic Pain
Keywords: pain self-management; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by recruitment clinic and dose of buprenorphine at enrollment (≤16 mg vs >16 mg) and randomized in 2x2 factorial design: 1) either to PSM or Usual Care, and then 2) either to POD or standard buprenorphine dosing. The randomization schema will be generated by the TREETOP Data Core using a stratified permuted block design and will be integrated into the web-based data collection and management system (REDCap).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual Care + Standard Buprenorphine Dosing (Active Comparator): Usual care, or "treatment as usual," refers to the standard of care that participants receive at their office-based addiction treatment (OBAT) clinic. This includes discussing issues related to chronic pain and opioid use (e.g., buprenorphine) with their provider and receiving clinical care for these conditions.
  Participants will continue standard buprenorphine or buprenorphine/naloxone dosing as part of normal clinical care.
  Interventions: Behavioral: Usual Care; Drug: Standard Buprenorphine Dosing Condition
- Usual Care + Patient-Oriented Dosing (POD) (Experimental): Usual care, or "treatment as usual," refers to the standard of care that participants receive at their office-based addiction treatment (OBAT) clinic. This includes discussing issues related to chronic pain and opioid use (e.g., buprenorphine) with their provider and receiving clinical care for these conditions.
  Patient-oriented dosing (POD) is a promising approach to using buprenorphine or buprenorphine/naloxone for treating participants with both opioid use disorder (OUD) and chronic pain. POD allows titration of buprenorphine or buprenorphine/naloxone dosing up to 32mg/day, split into four doses per day, based on the participant's pain level.
  Interventions: Drug: Patient-Oriented Dosing (POD); Behavioral: Usual Care
- Pain Self-Management (PSM) + Standard Buprenorphine Dosing (Experimental): Pain self-management (PSM) is a manualized behavioral intervention tailored for patients in outpatient-based addiction treatment (OBAT) programs. PSM consists of 12 intervention sessions, comprising 6 group sessions and 6 individual sessions.
  Participants will continue standard buprenorphine or buprenorphine/naloxone dosing as part of normal clinical care.
  Interventions: Behavioral: Pain Self-Management (PSM); Drug: Standard Buprenorphine Dosing Condition
- Pain Self-Management (PSM) + Patient-Oriented Dosing (POD) (Experimental): Pain self-management (PSM) is a manualized behavioral intervention tailored for patients in outpatient-based addiction treatment (OBAT) programs. PSM consists of 12 intervention sessions, comprising 6 group sessions and 6 individual sessions.
  Patient-oriented dosing (POD) is a promising approach to using buprenorphine or buprenorphine/naloxone for treating participants with both opioid use disorder (OUD) and chronic pain. POD allows titration of buprenorphine or buprenorphine/naloxone dosing up to 32mg/day, split into four doses per day, based on the participant's pain level.
  Interventions: Drug: Patient-Oriented Dosing (POD); Behavioral: Pain Self-Management (PSM)

INTERVENTIONS:
Drug: Patient-Oriented Dosing (POD) — Patient-oriented dosing (POD) is a promising approach to using buprenorphine or buprenorphine/naloxone to treat individuals with both OUD and chronic pain. It is based on existing evidence related to buprenorphine for the treatment of pain. POD allows participants to receive a daily dosage of bup up to 32mg/day, split up to 4 times per day.
  A response-guided dosing strategy, in which buprenorphine or buprenorphine/naloxone doses will be titrated based on a participant response, will be used to identify a dose regimen that is safe and effective. Due to inter-individual pharmacokinetic/pharmacodynamic variability, POD dosing will be individualized based on a participant's pain intensity and interference.
  Arms: Pain Self-Management (PSM) + Patient-Oriented Dosing (POD); Usual Care + Patient-Oriented Dosing (POD)
Behavioral: Pain Self-Management (PSM) — Pain self-management (PSM) is a manualized behavioral intervention consisting of 12 sessions, comprising 6 group and 6 individual sessions. The first session will be individual, followed by a group session, and then alternating weekly for the remainder of the intervention.
  Individual sessions will be led by a staff Interventionist trained in the pain self-management intervention. The interventionist will guide participants through a PSM study manual, providing education, teaching associated skills, and assisting with goal setting.
  Group sessions will be led by a Peer Facilitator who has experience with chronic pain, opioid use disorder, and buprenorphine treatment. These sessions will not have specific content but will serve as supportive forums for participants to discuss their experiences with the intervention, share tips for managing chronic pain, and provide mutual support.
  Arms: Pain Self-Management (PSM) + Patient-Oriented Dosing (POD); Pain Self-Management (PSM) + Standard Buprenorphine Dosing
Behavioral: Usual Care — Usual care, or "treatment as usual," refers to the standard of care that participants receive at their office-based addiction treatment (OBAT) clinic. This includes discussing issues related to chronic pain and opioid use (e.g., buprenorphine) with their provider and receiving clinical care for these conditions.
  Arms: Usual Care + Patient-Oriented Dosing (POD); Usual Care + Standard Buprenorphine Dosing
Drug: Standard Buprenorphine Dosing Condition — Participants will continue standard buprenorphine or buprenorphine/naloxone dosing as part of normal clinical care.
  Arms: Pain Self-Management (PSM) + Standard Buprenorphine Dosing; Usual Care + Standard Buprenorphine Dosing

SUMMARY:
This study seeks to improve the treatment of chronic pain in people who are taking buprenorphine (also known as Suboxone, Subutex, Zubsolv).

The research study is testing two different interventions along with usual clinical care:

1. Pain Self-Management (PSM): an educational program in which individuals with chronic pain work with a trained pain coach and a pain peer to explore strategies to effectively manage the daily problems that arise from chronic pain.
2. Patient-Oriented Dosing (POD): an alternative dosing of buprenorphine which will be adjusted based on pain levels.

The interventions will take place over a period of 12 weeks (3 months). Additionally, participants will complete surveys every 3 months for a period of 1 year (total of 5 survey visits). Participants will receive $50 compensation for each survey visit completed (up to $250 over one year) and can receive up to an additional $100 bonus compensation.

There are risks associated with participating in the study, including breach of confidentiality, psychological distress caused by discussing difficult topics, and risks associated with the POD intervention.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Adults at least 18 years old
2. Patient at a participating clinic
3. Ability to speak, read, and understand English
4. Capable of providing informed consent
5. Access to phone and/or internet
6. Documented diagnosis of Opioid Use Disorder (OUD)
7. On a stable dose of an oral or sublingual buprenorphine mono or combination product (<4 times per day, daily dosage <32 mg) for at least 7 days during incident new episode of care
8. Have high impact chronic pain (Grade 3), based on the Graded Chronic Pain Scale-Revised (GCPS-R)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Under 18 years of age
2. Have cancer-related pain
3. Are currently in jail, prison, or overnight facility as required by court of law or have pending legal action that could prevent participation in study activities
4. Currently prescribed 32mg of an oral or sublingual buprenorphine mono or combination product
5. Currently prescribed an injectable formulation of buprenorphine
6. Pregnancy or intention to become pregnant within 4 months of enrollment
7. Currently prescribed naltrexone or received naltrexone (Vivitrol) injection in the past 60 days
8. History of hypersensitivity to buprenorphine that a clinician-determined caused serious rash/hives/pruritus, bronchospasm, angioneurotic edema, or anaphylactic shock
9. Currently prescribed/taking methadone or have taken methadone in the past 30 days
10. Had an intentional suicide attempt within the past 3 months

Individuals with common comorbidities, such as depression, anxiety, or alcohol, methamphetamine, and other substance use disorders will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Interference as Assessed by the PROMIS SF v1.0 - Pain Interference 4a at 3 months Post-baseline | Baseline, 3 Months
  The PROMIS Pain Interference - Short Form 4a is a validated, self-report 4-item tool assessing pain interference over the past 7 days. The PROMIS SF v1.0 - Pain Interference 4a consists of 4 questions and uses a 5-point scale, ranging from 1 (not at all) to 5 (very much). The total raw score equals the sum the values of the response to each question. The raw score is converted to a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like pain interference, a T-score of 60 is one SD worse than average. That is, a person has more problems with pain hindering activities. By comparison, a pain interference T-score of 40 is one SD better than average.
  Change = 3 month score - baseline score

SECONDARY OUTCOMES:
Change from Baseline in Overall Pain as Assessed by the PEG at 3 months Post-baseline | Baseline, 3 Months
  The Pain, Enjoyment, and General Activity (PEG) Scale is a validated, self-report 3-item tool assessing pain intensity and interference over the past week. The PEG scale consists of 3 separate numerical scales. Each scale has ratings ranging from 0-10. The PEG score is calculated by averaging the three numbers; a higher score indicates greater pain.
  Change = 3 month score - baseline score
Change from Baseline in Pain Catastrophizing as Assessed by the Pain Catastrophizing Questionnaire-6-item at 3 months Post-baseline | Baseline, 3 Months
  The Pain Catastrophizing Scale is a validated, self-report 6-item tool assessing assess pain catastrophizing for chronic pain. The PCS-6 uses a 5-point scale, ranging from 0 (not at all) to 4 (all the time). The total score ranges from 0 to 24, with higher score representing greater catastrophic thinking.
  Change = 3 month score - baseline score
Proportion of Participants Retained in buprenorphine Treatment at 3 months Post-baseline | 3 Months
  Proportion retained is defined as # completed visits divided by # scheduled visits
Proportion of Participants Taking any MOUD at 3-, 6-, 9- and 12-months Post-baseline | 3 Months, 6 Months, 9 Months, 12 Months
  Measured by self-report and medical chart extraction
Change from Baseline in Self-efficacy as Assessed by the PROMIS Self-Efficacy for Managing Symptoms SF-4a at 3 months Post-baseline | Baseline, 3 Months
  The PROMIS Self-Efficacy for Managing Symptoms - Short Form 4a is a validated, self-report 4-item tool assessing current level of confidence to managing symptoms in relation to a chronic condition. The PROMIS SF v1.0 - Pain Interference 4a consists of 4 questions and uses a 5-point scale, ranging from 1 (I am not confident at all) to 5 ( I am very confident). The total raw score equals the sum the values of the response to each question. The raw score is converted to a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For example, a T-score of 55 on the PROMIS Self-Efficacy for Managing Emotions indicates that the respondent has greater self-efficacy for managing their emotions than the general chronic condition population (i.e., half a standard deviation higher).
  Change = 3 month score - baseline score
Number of Days Non-prescribed Opioids were Used in the past 30 days as Assessed by the Modified ASI at 3-months Post-baseline | 3 Months
  The modified ASI is a validated, self-report tool which includes questions from the Addiction Severity Index section on drug and alcohol use and includes questions about specific opioids used. The number of days in the last 30 that a participant reports using heroin, fentanyl, and/or opioid analgesics (percocet, oxycodone, oxycontin, vicodin, dilaudid, hydrocodone, hydromorphone, morphine, or codeine) will be summed for the outcome "Number of days non-prescribed opioids were used in the past 30 days." Number of days may range from 0 to 90.
Total score on the IMPOWR Opioid Misuse Screening scale at 3 months Post-baseline | 3 Months
  The IMPOWR Opioid Misuse Screening scale is an exploratory, self-report scale consisting of 4 questions about the use of prescribed pain medications. Each question response ranges from Never (0) to Almost Always (4) with a possible summed score ranging from 0 to 16, with higher scores indicating more severe misuse.

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Winstanley, PhD, Principal Investigator — University of Pittsburgh
Locations (13):
- United States (13):
  - Alcohol and Drug Abuse Program (ADAP) - UM Addiction Treatment Center, Baltimore, Maryland
  - MATClinics, Dundalk, Maryland
  - Wells House, Hagerstown, Maryland
  - Central City Concern (CCC), Portland, Oregon
  - Recovery Works Northwest (RWNW), Portland, Oregon
  - OHSU Harm Reduction Bridges to Care (HRBR), Portland, Oregon
  - OHSU Internal Medicine Clinic (IMC), Portland, Oregon
  - UPMC Latterman Family Health Center, McKeesport, Pennsylvania
  - UPMC St. Margaret Family Health Center, New Kensington, Pennsylvania
  - UPMC Magee-Womens Pregnancy and Women's Recovery Center (PWRC), Pittsburgh, Pennsylvania
  - UPMC Internal Medicine Recovery Engagement Program (IM-REP), Pittsburgh, Pennsylvania
  - WVU Crisis Support & Recovery Center, Martinsburg, West Virginia
  - WVU Chestnut Ridge Comprehensive Addiction Treatment Program (COAT), Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy) and data for this study will be available to the public through the IMPOWR Dissemination Education and Coordination Center (IDEA-CC) (https://heal.nih.gov/research/clinical-research/integrative-management-chronic-pain).
Supporting Information: Study Protocol, SAP
Time Frame: De-identified data will be made available within 18 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Access to trial IPD may be made available to individuals that submit a request along with the required documents to the IMPOWR data committee. Data access requires approval by the IMPOWR data committee and the individual must agree to comply with the data sharing policies of IMPOWR and HEAL.
URL: https://heal.nih.gov/research/clinical-research/integrative-management-chronic-pain